CLINICAL TRIAL: NCT04275739
Title: Episodic Future Thinking as a Brief Alcohol Intervention for Heavy Drinking College Students: A Pilot Feasibility Study
Brief Title: Brief Academic Future Thinking Intervention for College Student Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Principal Investigator, Andrew Voss, Principal Investigator, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-FY2017-587
Record Dates: First submitted 2020-02-05; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Heavy Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Episodic Future Thinking (Experimental)
  Interventions: Behavioral: Academic Episodic Future Thinking
- Control: Vivid Memory Task (Active Comparator)
  Interventions: Other: Vivid Memory Task

INTERVENTIONS:
Behavioral: Academic Episodic Future Thinking — Brief Academic goal related EFT intervention involving desirable outcomes of current academic goals
  Arms: Experimental: Episodic Future Thinking
Other: Vivid Memory Task — Matched for time control task involving recall of vivid memories of distinct events/actions from a children's story
  Arms: Control: Vivid Memory Task

SUMMARY:
The present study investigated the feasibility, acceptability, and initial utility of a brief academic goal-relevant episodic future thinking (A-EFT) task among heavy college drinkers.

First, the study attempts to extend the temporal reach of EFT interventions which have demonstrated immediate reductions in discounting, and alcohol demand. The current study utilized a longitudinal design to evaluate whether EFT can change drinking behavior outside the lab in heavy drinking college students. The two-group experimental design included an active control group, weekly booster contact, and 1-month follow-up. Second, this study seeks to investigate whether the process of engaging in EFT is sufficient to produce effects when cues are not presented during the decision-making task. Lastly, this study adds an academic goal-related focus to the EFT task based on previous research indicating that forming meaningful academic goals is protective against drinking and associated problems.

ELIGIBILITY:
Inclusion Criteria:

* Full-time Freshman/Sophomore Student
* 2+ Recent heavy drinking episodes (4/5 standard drinks in one sitting for men/women)

Exclusion Criteria:

* Current or past substance abuse treatment
* Current moderate/severe depressive symptoms

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Daily Drinking Questionnaire | Baseline
  Indicate how many standard drinks were consumed on each day of a "typical week" in the past month
Daily Drinking Questionnaire | 1-month post
  Indicate how many standard drinks were consumed on each day of a "typical week" in the past month
Alcohol-Related Consequences | Baseline
  Young Adult Alcohol Consequences Questionnaire - Indicate "yes" or "no" to experiencing each alcohol-related consequences in the past month
Alcohol-Related Consequences | 1-month post
  Young Adult Alcohol Consequences Questionnaire - Indicate "yes" or "no" to experiencing each alcohol-related consequences in the past month
Alcohol Demand | Baseline
  Alcohol Purchase Task - Indicate hypothetical alcohol purchase behavior at a variety of price points
Alcohol Demand | Post-session - immediately after intervention;control
  Alcohol Purchase Task - Indicate hypothetical alcohol purchase behavior at a variety of price points
Alcohol Demand | 1-month post
  Alcohol Purchase Task - Indicate hypothetical alcohol purchase behavior at a variety of price points
Delayed Reward Discounting | Baseline
  5-Choice Minute Discounting task - Indicate preference for various choices of immediate small vs. larger delayed rewards
Delayed Reward Discounting | Post-session - immediately after intervention/control
  5-Choice Minute Discounting task - Indicate preference for various choices of immediate small vs. larger delayed rewards
Delayed Reward Discounting | 1-month post
  5-Choice Minute Discounting task - Indicate preference for various choices of immediate small vs. larger delayed rewards

SECONDARY OUTCOMES:
Protective Behavioral Strategies | Baseline
  Indicate frequency of use of each protective strategy on a 1-6 Likert-type scale (1 = Never, 6 = Always)
Protective Behavioral Strategies | 1-month post
  Indicate frequency of use of each protective strategy on a 1-6 Likert-type scale (1 = Never, 6 = Always)
Academic Engagement | Baseline
  Single item assessing time spent studying during the past week
Academic Engagement | 1-month post
  Single item assessing time spent studying during the past week

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Memphis, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Voss AT, Jorgensen MK, Murphy JG. Episodic future thinking as a brief alcohol intervention for heavy drinking college students: A pilot feasibility study. Exp Clin Psychopharmacol. 2022 Jun;30(3):313-325. doi: 10.1037/pha0000451. Epub 2021 Feb 25. PMID 33630649